CLINICAL TRIAL: NCT02021058
Title: Effect of an Experimental Infant Formula in Unsettled Infants Experiencing Feeding Intolerance
Brief Title: Study in Unsettled Infants Experiencing Feeding Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13.10.INF
Record Dates: First submitted 2013-11-22; First posted 2013-12-27 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Feeding Disorder
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Formula (Experimental): Experimental Formula
  Interventions: Other: Experimental Formula
- Standard Formula (Other): Standard Control formula
  Interventions: Other: Standard control formula

INTERVENTIONS:
Other: Experimental Formula — Experimental formula
  Arms: Experimental Formula
Other: Standard control formula — Standard Infant formula
  Arms: Standard Formula

SUMMARY:
Multinational, multicenter, clinical trial. To evaluate the effect of an experimental formula on GI symptoms and associated behaviors in unsettled infants with parent-reported feeding intolerance

DETAILED DESCRIPTION:
The purpose of the present study is therefore to evaluate the effect of an experimental formula in an unsettled formula-fed infant population whose parents are considering switching formulas due to perceived feeding intolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Full term infants, singleton, healthy at birth
2. Infants of parent(s)/LAR who have previously made the decision to exclusively formula feed their infant.
3. Infants exclusively consuming a standard formula for a minimum of 3 consecutive days prior to enrolment.
4. Infant's parent(s)/LAR are of legal age of consent and are willing and able to fulfil the requirements of the study protocol.

Exclusion Criteria:

1. Infants who are consuming any amount of supplemental human milk
2. Infants who are consuming weaning foods or beverages other than infant formula
3. Infants with known cow's milk allergy or family history of siblings with documented cow's milk protein intolerance/allergy
4. Infants who have a medical condition or history that could cause or contribute to feeding intolerance
5. Infants who received any other investigational intervention or who have participated in another clinical trial prior to enrolment

Ages: 30 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 259 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to 14 days in fuss-cry behavior | from baseline to 14 days
  fuss-cry behavior per 24 hours

SECONDARY OUTCOMES:
Change from baseline to 14 days in GI symptoms | from baseline to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Boosba Vivatvakin, MD, Principal Investigator — Pediatric Department, Faculty of Medicine, Chulalongkorn University
Locations (6):
- The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong
- Asian Hospital and Medical Center, City of Muntinlupa, Philippines
- Taiwan (3):
  - Chang Gung Memorial Hospital - Linkou, Hsiang, Taoyan Hsien
  - Mackay Memorial Hospital - Tamsui, New Taipei City
  - Mackay Memorial Hospital - Taipei, Taipei
- King Chulalongkorn Memorial Hospital - Faculty of Medicine, Chulalongkorn University, Pratumwan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vivatvakin B, Estorninos E, Lien R, Lee HC, Hon KLE, Lebumfacil J, Cercamondi CI, Volger S. Clinical Response to Two Formulas in Infants with Parent-Reported Signs of Formula Intolerance: A Multi-Country, Double-Blind, Randomized Trial. Glob Pediatr Health. 2020 Sep 25;7:2333794X20954332. doi: 10.1177/2333794X20954332. eCollection 2020. PMID 33029552